CLINICAL TRIAL: NCT00190619
Title: Efficacy and Safety of Duloxetine Compared With Placebo in Subjects Electing Surgery for Severe Pure Genuine Stress Incontinence
Brief Title: Efficacy and Safety of Duloxetine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2624; F1J-MC-SBAM
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Urinary Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine
Drug: Placebo

SUMMARY:
The purpose of this study is to monitor the long term safety and efficacy of duloxetine in the treatment of severe pure genuine stress incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Female out patients.
* Have a diagnosis of pure genuine stress incontinence on urodynamic study performed within 6 months prior to study entry.

Exclusion Criteria:

* Use of monoamine oxidase inhibitors within 14 days prior to study entry or at any time during the study.
* Suffer from severe constipation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-05; Study Completion 2006-05

PRIMARY OUTCOMES:
Assess the efficacy of duloxetine versus placebo for in women who have decided to proceed toward surgery for severe pure genuine stress incontinence

SECONDARY OUTCOMES:
Change in the disease-specific quality of life instrument (Incontinence Quality of Life) scores from baseline to endpoint.
Compare the efficacy of duloxetine with that of placebo measured by: Patient Global Impression Improvement questionnaire, Symptoms Frequency & Bothersomeness Questionnaire, and percent change in weekly pad usage
Assess the efficacy of duloxetine measured by percent change in incontinence episode frequency and incontinence pad usage, and Patient Global Impression Improvement scores
Assess subject satisfaction with duloxetine compared with placebo as measured by Patient Satisfaction Questionnaire -2 (PSQ-2) and Patient Satisfaction Questionnaire - 4 (PSQ-4)
Compare the safety of duloxetine with that of placebo in the treatment of genuine stress incontinence based on vital signs, laboratory values, electrocardiogram findings, and the occurrence of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hrs, EST) or speak with your personal physician., London, United Kingdom